CLINICAL TRIAL: NCT06506552
Title: Inferior Mesenteric Artery Preservation in Laparoscopic Colorectal Resection for Diverticular Disease; Short and Long Term Effects in Defecatory Function
Brief Title: Effects of Inferior Mesenteric Artery Preservation in Laparoscopic Colorectal Resection for Diverticular Disease.
Acronym: EIMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, MD, PhD, FACS, Research fellow, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS-056
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Colonic Diverticuar Disease; Defecatory Functions; Fecal Incontinence; Constipation
Keywords: defecatory function; anterior resection syndrome; constipation; diverticular disease; fecal incontinence; fragmented evacuation
MeSH Terms: conditions — Fecal Incontinence; Constipation; Diverticular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior mesenteric artery preservation (Experimental): Performing colorectal resection for diverticular disease the IMA was preserved ligating the sigmoids arteries close to colonic wall.
  Interventions: Procedure: IMA preserving
- Inferior mesenteric ligation (Active Comparator): Performing colorectal resection the IMA was sectioned just below the origin of left colic artery.
  Interventions: Procedure: IMA sectioning

INTERVENTIONS:
Procedure: IMA preserving — Performing left hemicolectomy, sigmoidectomy or rectal resection the IMA was preserved ligating the sigmoids arteries close to the colonic wall
  Arms: Inferior mesenteric artery preservation
Procedure: IMA sectioning — Performing left emicolectomy, sigmoidectomy or rectal resection the IMA is sectioned after the origin of left colic artery.
  Arms: Inferior mesenteric ligation

SUMMARY:
This is a prospective randomized study aimed to verifying the short and long-term results of inferior mesenteric artery preservation following colorectal resection for diverticular disease

DETAILED DESCRIPTION:
This study wants to demonstrate that the preservation of the inferior mesenteric artery allow to improve postoperative defecatory function and improve patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35
* ASA I-III
* Hinchey I-III

Exclusion Criteria:

* BMI > 35
* ASA IV
* Hinchey IV
* Previous procedures that could have been modified the nervous mesenteric pattern (surgery, radiotherapy or chemotherapy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Defecatory disorders | 6 months from surgery
  the presence of defecatory disorders was evaluated (Costipation, Evacuation frequency,evacuation urgency, fragmented evacuation,flatus incontinence, liquid incontinence)
Defecatory disorders | 12 months from surgery
  the presence of defecatory disorders was evaluated (Costipation, Evacuation frequency,evacuation urgency, fragmented evacuation,flatus incontinence, liquid incontinence)
Defecatory disorders | 6 years from surgery
  the presence of defecatory disorders was evaluated (Costipation, Evacuation frequency,evacuation urgency, fragmented evacuation,flatus incontinence, liquid incontinence)

SECONDARY OUTCOMES:
Constipation | 6 months from surgery
  The incidence and severity of postoperative constipation was evaluated with Cleveland Clinic Constipation Score ( score range from 0 to 30, the higher score defines worse constipation status)
Constipation | 12 months from surgery
  The incidence and severity of postoperative constipation was evaluated with Cleveland Clinic Constipation Score ( score range from 0 to 30, the higher score defines worse constipation status)
Constipation | 6 years from surgery
  The incidence and severity of postoperative constipation was evaluated with Cleveland Clinic Constipation Score ( score range from 0 to 30, the higher score defines worse constipation status)
Incontinence | 6 months from surgery
  The presence of fecal incontinence was evaluated with Cleveland Clinic Incontinence Score( score range from 0 to 20, the higher score defines worse symptoms)
Incontinence | 12 months from surgery
  The presence of fecal incontinence was evaluated with Cleveland Clinic Incontinence Score( score range from 0 to 20, the higher score defines worse symptoms)
Incontinence | 6 years from surgery
  The presence of fecal incontinence was evaluated with Cleveland Clinic Incontinence Score( score ranges from 0 to 20, the higher score defines worse symptoms)
Anorectal Muscles function | 6 months from surgery
  The anorectal muscles function was evaluated with anorectal manometry( sphincter lenght, maximum squeeze pression, resting anal pressure, squeeze duration, maximum pressure sustained)
Anorectal Muscles function | 6 years from surgery
  the anorectal muscles function was evaluated with anorectal manometry ( sphincter lenght, maximum squeeze pression, resting anal pressure, squeeze duration, maximum pressure sustained)
Postoperative quality of life | 6 months from surgery
  the postoperative QOL(quality of life) was evaluated with EORTC-30 tests( European organization for research and treatment of cancer, scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms)
Postoperative quality of life | 12 months from surgery
  the postoperative QOL was evaluated with EORTC-30 tests( European organization for research and treatment of cancer,scores range from 0 to 100; a higher score represents a higher "better" level of functioning, or a higher "worse" level of symptoms
Postoperative quality of life | 6 years from surgery
  The postoperative QOL was evaluated with EORTC-30 tests( European organization for research and treatment of cancer,scores range from 0 to 100; a higher score represents a higher "better" level of functioning, or a higher "worse" level of symptoms)
Postoperative quality of life | 12 months from surgery
  The postoperative QOL was evaluated with EORTC-29 tests (European organization for research and treatment of cancer each question goes from 1 to 4 , the higher score defines worse symptoms)
Postoperative quality of life | 6 years from surgery
  The postoperative QOL was evaluated with EORTC-29 tests (European organization for research and treatment of cancer each question goes from 1 to 4 , the higher score defines worse symptoms)
Postoperative quality of life | 6 months from surgery
  The postoperative QOL was evaluated with EORTC-29 tests (European organization for research and treatment of cancer each question goes from 1 to 4 , the higher score defines worse symptoms)
Postoperative quality of life | 6 months from surgery
  The postoperative QOL(quality of life) was evaluated with SF-36 score (Short form-36 score, each item scored from 0 to 100, the higher scores defines a favorable health state)
Postoperative quality of life | 12 months from surgery
  The postoperative QOL was evaluated with SF-36 score (Short form-36 score, each item scored from 0 to 100, the higher scores defines a favorable health state)
Postoperative quality of life | 6 years from surgery
  The postoperative QOL was evaluated with SF-36 score (Short form-36 score, each item scored from 0 to 100, the higher scores defines a favorable health state)
Postoperative surgical complication | 1 month from surgery
  The incidence of postoperative surgical complications was evaluated

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mari FS, Chiarini L, Trampetti L, Savina C, Cosmi F, Cicolani A, Gasparrini M, Brescia A. Preservation of inferior mesenteric artery reduces short- and long-term defecatory dysfunction after laparoscopic colorectal resection for diverticular disease: An RCT. Surg Endosc. 2025 Mar;39(3):1761-1769. doi: 10.1007/s00464-024-11490-7. Epub 2025 Jan 15. PMID 39814952